CLINICAL TRIAL: NCT04378426
Title: Nitrous Oxide for Posttraumatic Stress Disorder (PTSD): A Phase IIa Trial
Brief Title: Nitrous Oxide for PTSD
Acronym: N2OP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Use of VA hospital research space is indefinitely delayed due to prioritization of clinical cases delayed by COVID
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MHBB-009-19S; I01CX001789 (NIH); 53017 (Other: IRB)
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Results first posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: PTSD
Keywords: PTSD; Nitrous Oxide
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Nitrous Oxide; Midazolam; Nitrogen; Oxygen; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled clinical trial including two groups: Experimental (admixture of up to 50% nitrous oxide and 50% oxygen plus IV saline) and Active Comparator (admixture of up to 50% nitrogen and 50% oxygen plus 0.045mg/kg midazolam).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinding Protections: First, the investigators will separate personnel and location of the team providing study drug from the team performing psychiatric evaluations. Independent evaluators (IEs) blind to treatment assignment will assess participants . Second, records for drug administration will be kept separate from psychiatric assessment case report forms until completion of the study. Third, all participants will be blinded as to the nature of the inhaled gas and IV drug at each session; all participants will be informed that they will receive either nitrous oxide and IV saline or an air mixture with a high nitrogen component and IV midazolam. Integrity of the blinding will be assessed by recording each patient's guess as to which drug was received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nitrous Oxide (Experimental): PTSD participants in this arm will receive and admixture of up to 50%nitrous oxide and 50% oxygen plus intravenous saline
  Interventions: Drug: Nitrous Oxide; Drug: Oxygen; Drug: Saline
- Midazolam (Active Comparator): PTSD participants in this arm will receive and admixture of up to 50%nitrogen and 50% oxygen plus intravenous 0.045mg/kg midazolam
  Interventions: Drug: Midazolam; Drug: Nitrogen; Drug: Oxygen

INTERVENTIONS:
Drug: Nitrous Oxide — PTSD participants in this arm will receive and admixture of up to 50% nitrous oxide and 50% oxygen plus intravenous saline
  Arms: Nitrous Oxide
Drug: Midazolam — PTSD participants in this arm will receive and admixture of up to 50%nitrogen and 50% oxygen plus intravenous 0.045mg/kg midazolam
  Arms: Midazolam
Drug: Nitrogen — PTSD participants in this arm will receive and admixture of up to 50%nitrogen and 50% oxygen plus intravenous 0.045mg/kg midazolam
  Arms: Midazolam
Drug: Oxygen — inhaled gas
Drug: Saline — Placebo infusion
  Arms: Nitrous Oxide

SUMMARY:
Post-traumatic stress disorder (PTSD) seriously disrupts the lives of many Veterans. Current first-line treatments, serotonin reuptake inhibitors or prolonged exposure therapy, take weeks to months to bring meaningful improvement, leaving Veterans experiencing prolonged suffering. A promising new treatment approach for rapidly reducing PTSD symptoms is nitrous oxide, an inhalation anesthetic and putative glutamate modulator that diminishes depression symptoms within 1 day and has limited side effects. If shown to be similarly effective in PTSD, nitrous oxide may add dramatically to the treatment armamentarium by bringing rapid symptom decrease before longer-term therapies take hold. The proposed projects test the efficacy of nitrous oxide in relieving Veteran's PTSD symptoms and, in parallel, explore how nitrous oxide may modify cognitive and pain outcomes.

DETAILED DESCRIPTION:
The proposed projects will examine the efficacy of nitrous oxide in relieving Veteran's PTSD symptoms and in parallel, explore whether nitrous oxide improves cognitive and pain outcomes. Specifically, the investigators will first assess whether nitrous oxide treatment improves PTSD symptoms within 1 week. In parallel, the investigators will explore whether the treatment improves co-existing depression and pain. In addition, the investigators will explore nitrous oxide's effects on a PTSD-associated impairment that is often overlooked - disruption in cognitive control, a core neurobiological process critical for regulating thoughts and for successful daily functioning.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* primary diagnosis of PTSD
* sufficient severity of PTSD symptoms
* capacity to provide informed consent

Exclusion Criteria:

* psychiatric or medical conditions that make participation unsafe
* pregnant or nursing females
* concurrent use of any medications that might increase the risk of participation (e.g. drug interactions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn I Rodriguez, MD PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
No data will be shared without approval of sponsor and IRB.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nitrous Oxide | Midazolam
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study discontinued due to unsufficient space due to backlog of clinical patients due to COVID
Groups:
- Total: Total of all reporting groups
Arm/Group | Nitrous Oxide | Midazolam | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (0) |  | 49 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 1 |  | 1
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 1 |  | 1
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 0 |  | 0
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1
CAPS 5 [Mean (Standard Deviation); unit: units on a scale] — For the CAPS-5 the minimum units are 0 and maximum units are 80. The higher the number on the CAPS-5, the more severe the PTSD symptoms.
  units on a scale | 64 (0) |  | 64 (0)

OUTCOME MEASURES:

1. Primary Outcome: Improvement in the Severity of PTSD as Measured by the Clinician Administered PTSD Scale DSM5 (CAPS-5)
Description: Improvement in PTSD severity is measured by the Clinician Administered PTSD Scale DSM-5 (CAPS-5). It measures frequency and intensity of PTSD-related symptoms. For the CAPS-5 the minimum units are 0 and maximum units are 80. The higher the number on the CAPS-5, the more severe the PTSD symptoms. Response is defined as a change in the CAPS-5 of at least 12 points, which represents meaningful improvement in clinical PTSD symptoms.
Time Frame: 1 week
Population: The study was terminated in partnership with program officer given that the nitrous oxide administration space in the hospital (which had been used pre-pandemic) is longer available - it is being used exclusively for clinical care to keep up with the clinical backlog of cases due to the pandemic. This delay will continue for the foreseeable future. COVID-19 has had far-reaching impact on the feasibility of the study, which will not meet its recruitment goal in the foreseeable future.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nitrous Oxide | Midazolam
Number analyzed (Participants) | 1 | 0
units on a scale | 46 (0) |

ADVERSE EVENTS:
Time Frame: 1 week
Description: Only 1 participant was recruited before the study was terminated.
Arm/Group | Nitrous Oxide | Midazolam
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nitrous Oxide (N=1) | Midazolam (N=0)
nausea (Gastrointestinal disorders) | 1 | NA
dizziness (Nervous system disorders) | 1 | NA
poor coordination (Nervous system disorders) | 1 | NA
poor concentration (Nervous system disorders) | 1 | NA
fatigue (Nervous system disorders) | 1 | NA
general malaise (Nervous system disorders) | 1 | NA
tingling in toes (Nervous system disorders) | 1 | NA

LIMITATIONS AND CAVEATS:
The study was terminated in partnership with program officer given that the nitrous oxide administration space in the hospital (which had been used pre-pandemic) is longer available - it is being used exclusively for clinical care to keep up with the clinical backlog of cases due to the pandemic. This delay will continue for the foreseeable future. COVID-19 has had far-reaching impact on the feasibility of the study, which will not meet its recruitment goal in the foreseeable future.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/26/NCT04378426/Prot_002.pdf
  • Statistical Analysis Plan (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/26/NCT04378426/SAP_003.pdf